CLINICAL TRIAL: NCT04185220
Title: Phase 1 Study of Recombinant Human IL-15 (rhIL-15) and Mogamulizumab for Patients With Refractory or Relapsed Adult T-Cell Leukemia and Mycosis Fungoides/Sezary Syndrome
Brief Title: Phase I Study of Recombinant Human IL-15 (rhIL-15) and Mogamulizumab for People With Refractory or Relapsed Adult T-Cell Leukemia and Mycosis Fungoides/Sezary Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200011; 20-C-0011
Record Dates: First submitted 2019-12-03; First posted 2019-12-04 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Adult T-Cell Lymphoma/Leukemia; Sezary Syndrome; Mycosis Fungoides
Keywords: Antibody-Dependent Cell Cytotoxicity (ADCC); CCR4; Monoclonal Antibody
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Sezary Syndrome; Mycosis Fungoides | interventions — Interleukin-15; IL15RA protein, human; mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1- Experimental Treatment: Dose Escalation (Experimental): Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at escalating doses of 2 and 4 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kgdays 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle to determine MTD.
  Interventions: Drug: Recombinant human Interleukin-15 (rhIL-15); Biological: Mogamulizumab
- 2- Experimental Treatment: Dose Expansion (Experimental): Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at the maximum tolerated dose (MTD) on days 1- 5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kgdays 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle.
  Interventions: Drug: Recombinant human Interleukin-15 (rhIL-15); Biological: Mogamulizumab

INTERVENTIONS:
Drug: Recombinant human Interleukin-15 (rhIL-15) — Interleukin 15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation 3 + 3 system with a starting dose of 2 mcg/kg/day and a second dose level of 4 mcg/kg/day on days 1-5 of each of six cycles.
  Other Names: Human interleukin 15
Biological: Mogamulizumab — Mogamulizumab (intravenous (IV) over at least 1 hour) will be administered at a dose of 1 mg/kg on days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle. Treatment will continue for a maximum of 6 cycles.
  Other Names: Poteligeo

SUMMARY:
Background:

Adult T-cell leukemia/lymphoma (ATLL) and mycosis fungoides/Sezary syndrome (MF/SS) are cancers that form in the T cells, a type of white blood cell that helps with the body's immune response. A combination of drugs might be able to better treat these cancers than existing therapies.

Objective:

To test if the drugs interleukin-15 (IL-15) and mogamulizumab are safe and effective to treat people with Adult T-Cell Leukemia and Mycosis Fungoides/Sezary Syndrome (ATLL or MF/SS).

Eligibility:

People ages 18 and older with relapsed ATLL or MF/SS that has not responded to at least one standard treatment

Design:

Participants will be screened with:

Medical history

Physical exam

Blood (including human immunodeficiency virus (HIV), hepatitis B and C), urine, lung, and heart tests

Bone marrow tests (if needed): A needle inserted in the participants hip will take a small amount of marrow.

Computed tomography (CT), positron emission tomography (PET) and/or magnetic resonance imaging (MRI) scans

Tumor biopsy (if needed): A needle will take out a small piece of the participants tumor.

Participants will get the study drugs by vein for up to six 28-day cycles. They will get IL-15 the first 5 days of each cycle. They will get mogamulizumab on days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of the other cycles. They will be hospitalized for 1 week in cycle 1. They may need to get a midline catheter. This is a soft tube put into a vein leading to the heart.

Participants will have repeats of the screening tests throughout the study.

After treatment, participants will have visits every 60 days for 6 months, every 90 days for 2 years, and then every 6 months for 2 years.

DETAILED DESCRIPTION:
Background:

* Advanced mycosis fungoides, its leukemic form Sezary syndrome (MF/SS), and adult T- cell leukemia/lymphoma (ATLL) are all aggressive mature T-cell malignancies which are considered incurable without an allogeneic stem cell transplant.
* Mogamulizumab is a defucosylated monoclonal antibody directed towards C-C Motif Chemokine Receptor 4 (CCR4), a chemokine receptor expressed by the majority of MS/SS and ATLL cells. It is approved by the United States Food and Drug Administration for treatment of relapsed MF/SS and is recommended by the National Comprehensive Cancer Network for treatment of ATLL.
* Defucosylation of mogamulizumab is thought to enhance its capacity for antibody- dependent cell cytotoxicity (ADCC), which is mediated by natural killer (NK) cells and macrophages.
* The immunologic effects of recombinant human Interleukin-15 (rhIL-15), a stimulatory cytokine that promotes the differentiation and activation of natural killer (NK) cells, monocytes and long- term cluster of differentiation 8 (CD) 8+ memory T-cells, has been assessed in several phase I trials in cancer patients.
* Concomitant administration of rhIL-15 with mogamulizumab may further enhance the ADCC capacity of the antibody and result in improved efficacy for patients with CCR4- expressing cancers.

Objectives:

-To determine the safety and toxicity profile and the maximum tolerated dose (MTD) of continuous intravenous infusion (civ) rhIL-15 administration in combination with standard intravenous (IV) mogamulizumab treatment

Eligibility:

* Age greater than or equal to 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1
* Histologically or cytologically confirmed mycosis fungoides/S(SqrRoot)(Copyright)zary syndrome or adult T- cell leukemia/lymphoma relapsed after or refractory to at least one line of systemic treatment.
* Adequate organ and marrow function

Design:

* Open-label, single-center, non-randomized phase I study
* Standard "3 + 3" design will be used to determine the maximum tolerated dose (MTD) of dose-escalated recombinant human Interleukin-15 (rhIL-15) with fixed dose of mogamulizumab, with an expansion cohort at the MTD
* Maximum 6 cycles (28-day cycles) of combination therapy
* To explore all dose levels, including further evaluation in a dose expansion cohort, and to account for unevaluable patients the accrual ceiling will be set at 20 patients.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have one of the following histologically or cytologically proven relapsed and/or refractory to at least one line of systemic treatment, T-cell malignancies confirmed by the Laboratory of Pathology, National Cancer Institute (NCI): mycosis fungoides/Sezary syndrome, or adult T-cell leukemia (chronic, acute, or lymphoma subtype by Shimoyama criteria)
2. Patients with luster of differentiation 30 (CD30)+ Mycosis Fungoides/Sezary Syndrome (MF/SS) must have relapsed after or become intolerant to treatment with brentuximab vedotin
3. A formalin fixed tissue block or 15 slides of tumor sample (archival or fresh) must be available for performance of correlative studies. NOTE: Patients must be willing to have a tumor biopsy if prior tissue or adequate archival tissue is not available (i.e., post- enrollment and prior to treatment).
4. Disease must be measurable with at least one measurable lesion by Response Evaluation Criteria in Lymphoma (RECIL 2017) or modified severity-weighted assessment tool (mSWAT) criteria, or have an abnormal clonal T-cell population detectable by peripheral blood flow cytometry
5. Age >18 years

   NOTE: Because no dosing or adverse event data are currently available on the use of rhIL-15 in combination with mogamulizumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 80%
7. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count: greater than or equal to 1,000/mcL
   * Platelets: > 100,000/mcL
   * Total bilirubin: less than or equal to 1.5 X institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)Serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT)Serum glutamic pyruvic transaminase (SGPT): less than or equal to 2.5 X institutional ULN
   * Serum creatinine: less than or equal to 1.5 X institutional ULN, OR Creatinine clearance: greater than or equal to 50 mL/min/1.73 m2 for patients with creatinine levels >1.5 institutional ULN
8. Negative serum or urine pregnancy test at screening for women of childbearing potential (WOCBP)

   NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of rhIL-15 and mogamulizumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

1. Patients with other T-cell leukemias/lymphomas not specified in the inclusion criteria
2. Anti-cancer treatment within 2 weeks of the first dose of rhIL-15 and mogamulizumab (4 weeks for anti-cancer monoclonal antibody or investigational agents, 6 weeks for donor lymphocyte infusion,100 days for allogeneic stem cell transplant)
3. Systemic treatment for acute or chronic graft versus host disease (GVHD) within 12 weeks of the first dose of rhIL-15 and mogamulizumab
4. Cohort 1 (Dose Escalation) only: history of grade 3/4 GVHD, or active grade 1/2 GVHD regardless of treatment
5. Persisting toxicity related to prior therapy of grade > 1, with the exception of the following: alopecia, sensory neuropathy grade less than or equal to 2, or other grade less than or equal to 2 not constituting a safety risk based on investigator's judgment
6. Patients who are receiving any other investigational agents
7. Current use of immunosuppressive medication, EXCEPT for the following:

   * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
   * Systemic corticosteroids at physiologic doses less than or equal to 10 mg/day of prednisone or equivalent; or,
   * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication)
8. Patients with previous malignant disease other than the target malignancy within the last 3 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ
9. Cohort 1 (Dose Escalation) only: Active or history of any autoimmune disease thought to be unrelated to their malignancy; for Cohort 2 (Dose Expansion), patients with history of autoimmune disease who are not on active immunosuppressive therapy
10. Patients with asthma requiring chronic inhaled or oral corticosteroids, or history of asthma requiring mechanical ventilation. Patients with a history of mild asthma that are on or can be switched to non-corticosteroid bronchodilator regimens are eligible
11. Patients with active bacterial infections, documented human immunodeficiency virus (HIV) infection or positive HIV 1/2 antibodies at screening, polymerase chain reaction (PCR) evidence for active or chronic hepatitis B or hepatitis C, or positive screening hepatitis B virus (HBV)/hepatitis C virus (HCV) serology without documentation of successful curative treatment
12. Presence of uncontrolled intercurrent illnesses including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cognitive impairment, active substance abuse, or psychiatric illness/social situations that in the view of the Investigator would preclude safe treatment and limit compliance with study requirements
13. Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding. Because there is no significant preclinical information regarding the risks to a fetus or a newborn infant, all pregnant or breastfeeding woman will be excluded from participation in this trial
14. History of allergic reactions attributed to compounds of similar chemical or biologic composition to rhIL-15 or mogamulizumab, unless felt to be in the best interests of the patient in the opinion of the investigator
15. Patients who received a live vaccine within 30 days of planned start of study therapy. Vaccination with a live vaccine while on trial is prohibited. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milos Miljkovic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon MJ, Dubois S, Miljkovic MD, Ng S, Bryant B, Lakhotia R, Melani C, Pittaluga S, Conlon K, Waldmann T, Staudt LM, Wilson WH, Roschewski M. A phase 1 study of interleukin-15 in combination with mogamulizumab in relapsed and refractory T-cell malignancies. Blood Neoplasia. 2024 Nov 2;2(1):100054. doi: 10.1016/j.bneo.2024.100054. eCollection 2025 Feb. PMID 40546724
- [Derived] Dubois SP, Miljkovic MD, Fleisher TA, Pittaluga S, Hsu-Albert J, Bryant BR, Petrus MN, Perera LP, Muller JR, Shih JH, Waldmann TA, Conlon KC. Short-course IL-15 given as a continuous infusion led to a massive expansion of effective NK cells: implications for combination therapy with antitumor antibodies. J Immunother Cancer. 2021 Apr;9(4):e002193. doi: 10.1136/jitc-2020-002193. PMID 33883258
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0011.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Interleukin-15 2mcg/kg/Day): Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at 2 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kg days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle to determine MTD.
- Dose Level 2 (Interleukin-15 4mcg/kg/Day): Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at 4 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kg days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle to determine MTD.
Period: Dose Escalation
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Started | 3 | 3
Completed | 3 | 1
Not Completed | 0 | 2
Not completed — Stopped treatment early due to progressive disease, dose limiting toxicity and acute renal failure | 0 | 1
Not completed — Stopped treatment early on cycle 1/day 2 due to Gr 2 infusion reaction & resulting Gr 3 hip fracture | 0 | 1
Period: Dose Expansion
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.73) | 45.07 (14.04) | 52.13 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Recombinant Human Interleukin 15 (IL-15) (rhIL-15)
Description: The MTD is the dose level at which no more than 1 of up to 6 patients experience DLT during the DLT evaluation window(s), or the dose below that at which at least 2 (of ≤6) patients have DLT. A dose-limiting toxicity (DLT) is defined as: any grade 3, 4, or 5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably or definitely related to IL-15 or mogamulizumab.
Time Frame: 28 days
Measure: Number; unit: mcg/kg/day
Groups:
- All Participants: All participants that received Dose Level 1: Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at 2 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kg days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 and Dose Level 2: Interleukin-15 (IL-15) by continuous intravenous (CIV) infusion at 4 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with mogamulizumab by intravenous (IV) infusion at a dose of 1 mg/kg days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent cycle to determine MTD.
Arm/Group | All Participants
Number analyzed (Participants) | 6
mcg/kg/day | 2

2. Primary Outcome: Number of Grade 1-4 Treatment Related Adverse Events
Description: Adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 25 days for dose level 1, and 4 months and 14 days for dose level 2.
Measure: Number; unit: adverse events
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
adverse events
  Grade 1 Alanine aminotransferase increased | 2 | 1
  Grade 1 Aspartate aminotransferase increased | 2 | 1
  Grade 1 Bronchial infection | 1 | 0
  Grade 1 Chills | 1 | 0
  Grade 1 Diarrhea | 1 | 0
  Grade 1 Dysgeusia | 2 | 0
  Grade 1 Fatigue | 2 | 0
  Grade 1 Fever | 9 | 1
  Grade 1 Hypomagnesemia | 5 | 0
  Grade 1 Neutrophil count decreased | 1 | 1
  Grade 1 Rash maculo-papular | 3 | 0
  Grade 2 Alanine aminotransferase | 1 | 0
  Grade 2 Anemia | 9 | 0
  Grade 2 Aspartate aminotransferase | 2 | 0
  Grade 2 Capillary leak syndrome | 1 | 0
  Grade 2 Bronchial infection | 1 | 0
  Grade 2 Chills | 1 | 0
  Grade 2 Creatine phosphokinase increased | 1 | 0
  Grade 2 Diarrhea | 1 | 0
  Grade 2 Dysgeusia | 1 | 0
  Grade 2 Fatigue | 1 | 1
  Grade 2 Fever | 2 | 0
  Grade 2 Infusion related reaction | 1 | 1
  Grade 2 Neutrophil count decreased | 1 | 1
  Grade 2 Rash maculo-papular | 0 | 1
  Grade 3 Alanine aminotransferase | 1 | 0
  Grade 3 Anemia | 9 | 0
  Grade 3 Creatine phosphokinase increased | 2 | 0
  Grade 3 Fall | 0 | 1
  Grade 3 Hip fracture | 0 | 1
  Grade 3 Hypoalbuminemia | 2 | 0
  Grade 3 Infusion related reaction | 0 | 1
  Grade 3 Rash maculo-papular | 1 | 0
  Grade 4 Acidosis | 0 | 1
  Grade 4 Capillary leak syndrome | 0 | 1
  Grade 4 Creatine phosphokinase increased | 2 | 0
  Grade 4 Acute kidney injury | 0 | 1

3. Secondary Outcome: Event Free Survival
Description: Event-free survival (EFS) is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), or death, whichever occurs first.
Time Frame: Up to one year
Measure: Mean (Standard Error); unit: Months
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
Months | 4.2 (1.46) | 2.1 (0.63)

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first. Progressive Disease (PD) is new or increased lesions.
Time Frame: Up to one year
Measure: Mean (Standard Error); unit: Months
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
Months | 4.2 (1.46) | 2.1 (0.63)

5. Secondary Outcome: Number of Participants Overall Response
Description: Overall response was assessed by the Response Criteria for Adult T-cell Leukemia-Lymphoma. The response rate was determined and reported along with a 95% confidence interval. Complete Response (CR) is disappearance of all disease. Unconfirmed Complete Response (CRu) is stable residual mass in bulky lesion. Partial Response (PR) is regression of disease. Relapsed Disease (RD)/Progressive Disease (PD) is new or increased lesions. And Stable Disease (SD) is failure to attain CR/PR and no PD.
Time Frame: 6 cycles (one cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 0
  Relapsed Disease/Progressive Disease | 2 | 3
  Stable Disease | 0 | 0
  Unconfirmed Complete Response | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

7. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT) Possibly, Probably or Definitely Related to Interleukin 15 (IL-15) or Mogamulizumab.
Description: A DLT is defined as any grade 3 (severe), 4 (life-threatening), or 5 (death related to adverse event) toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably or definitely related to IL-15 or mogamulizumab.
Time Frame: First cycle of treatment (28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
Number analyzed (Participants) | 3 | 3
Participants
  Possibly related to Interleukin 15 | 0 | 0
  Probably related to Interleukin 15 | 0 | 0
  Definitely related to Interleukin 15 | 0 | 2
  Possibly related to mogamulizumab | 0 | 0
  Probably related to mogamulizumab | 0 | 0
  Definitely related to mogamulizumab | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 5 months and 25 days for dose level 1, and 4 months and 14 days for dose level 2.
Arm/Group | Dose Level 1 (Interleukin-15 2mcg/kg/Day) | Dose Level 2 (Interleukin-15 4mcg/kg/Day)
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Interleukin-15 2mcg/kg/Day) (N=3) | Dose Level 2 (Interleukin-15 4mcg/kg/Day) (N=3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Multi organ failure (General disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Interleukin-15 2mcg/kg/Day) (N=3) | Dose Level 2 (Interleukin-15 4mcg/kg/Day) (N=3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (18) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (2) | 0 (0)
CPK increased (Investigations) | 1 (4) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1)
Fever (General disorders) | 3 (13) | 1 (1)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Uric Acid increased (Renal and urinary disorders) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Oral ulcer Right upper lip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04185220/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT04185220/ICF_001.pdf